CLINICAL TRIAL: NCT01651130
Title: Carbetocin at Elective Cesarean Deliveries: A Dose-finding Study Part 3
Brief Title: Carbetocin at Elective Cesarean Delivery Part 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-04
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Postpartum Hemorrhage
Keywords: pregnancy; postpartum hemorrhage; Cesarean delivery; carbetocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Carbetocin 100mcg (Active Comparator): Carbetocin 100mcg, once following delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 20mcg (Active Comparator): Carbetocin 20mcg, once following delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 15mcg (Active Comparator): Carbetocin 15mcg, once following delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 10mcg (Active Comparator): Carbetocin 10mcg, following delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 5mcg (Active Comparator): Carbetocin 5mcg, following delivery of the fetal head.
  Interventions: Drug: Carbetocin
- Carbetocin 2mcg (Active Comparator): Carbetocin 2mcg, following delivery of the fetal head.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — Carbetocin IV, over 1 minute following delivery of the fetal head. Doses: 2, 5, 10, 15, 20 or 100mcg
  Other Names: Duratocin

SUMMARY:
Post-partum hemorrhage (PPH) is a major cause of maternal death worldwide. Oxytocin is the most common uterotonic drug used to prevent and treat PPH in North America, however, there are some limitations to its use. Oxytocin has a very short duration of action, which requires a continuous infusion to achieve sustained uterotonic activity. The Society of Obstetricians and Gynecologists of Canada (SOGC) has recently recommended a single 100mcg dose of carbetocin at elective Cesarean delivery to promote uterine contraction and prevent post partum hemorrhage (PPH), in lieu of the more traditional oxytocin regimens. Carbetocin lasts 4 to 7 times longer than oxytocin, with a similar side effect profile and apparent greater efficacy rate. However, a dose response study to determine the minimum effective dose of carbetocin has not yet been published. The investigators hypothesize that the minimum effective dose (ED90) is at least 20mcgs (or perhaps below) in women undergoing elective Cesarean delivery.

DETAILED DESCRIPTION:
The Society of Obstetricians and Gynecologists of Canada (SOGC) recently recommended a 100mcg intravenous bolus dose of carbetocin following Cesarean delivery.

Studies thus far show that carbetocin may be just as effective as oxytocin in promoting uterine contraction, with a similar side effect profile. In addition, patients receiving carbetocin may experience less blood loss, and require less additional uterotonics when compared with oxytocin. Two dose response studies conducted at our institution (by Cordovani et al, and Anandakrishnan et al) suggested no difference in efficacy of uterine contraction for doses of carbetocin between 20-120mcg. Hypotension was noted for all dose groups studied.

This study will be conducted as a prospective, randomized, up-down sequential allocation trial. The success or fail of a patient in the study will determine the dose given to future patients. Dosage will be increased for patients following a failed case, and kept the same for patients following successful cases. Following a successful case, there is also a 1 in 9 chance that the dose will be decreased for the next patient.

The results of this follow-up study will define the minimum required dose of carbetocin for uterine contraction, thus minimizing unnecessary side effects, improving quality and safety of patient care. It may also contribute in establishing carbetocin as a substitute to oxytocin for elective cesarean section at our institution as well as others.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for elective cesarean delivery under spinal anesthesia
* Patients who give written informed consent to participate

Exclusion Criteria:

* Patients who refuse to give written informed consent
* Patients who claim allergy or hypersensitivity to carbetocin or oxytocin
* Patients with conditions that predispose to uterine atony and postpartum hemorrhage such as placenta previa, multiple gestation, preeclampsia, eclampsia, macrosomia, polyhydramnios, uterine fibroids, previous history of uterine atony and postpartum bleeding, or bleeding diathesis.
* Patients with hepatic, renal, and vascular disease
* Patients requiring general anesthesia prior to the administration of the study drug.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Uterine tone | 2 minutes
  The obstetrician will assess uterine tone by palpation. Uterine tone will be rated as satisfactory (firm) or unsatisfactory (boggy). Unsatisfactory uterine tone will be treated with oxytocin as per the obstetrician.

SECONDARY OUTCOMES:
Uterine tone | 2 hours
  Uterine tone will be assessed by palpation 2 hours post-delivery by the nurse/obstetrician in the recovery room.
Blood loss | 48 hours
  Blood loss will be calculated through the difference in hematocrit values assessed prior to and at the end of 48 hours after the cesarean section.
Side effects | 2 hours
  Any of the following will be noted up to 2 hours post delivery: systolic blood pressure < 80% of pre-delivery values, tachycardia > 30% pre-delivery levels, bradycardia < 30% pre-delivery levels, other dysrhythmias, nausea, vomiting, chest pain, shortness of breath, headache, flushing, others

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Khan M, Balki M, Ahmed I, Farine D, Seaward G, Carvalho JC. Carbetocin at elective Cesarean delivery: a sequential allocation trial to determine the minimum effective dose. Can J Anaesth. 2014 Mar;61(3):242-8. doi: 10.1007/s12630-013-0082-9. Epub 2013 Nov 27. PMID 24281981